CLINICAL TRIAL: NCT05348187
Title: An Interventional, Prospective Clinical Performance Study Protocol, for the Testing of DNA Extracted From Tumor Tissue Biopsy Samples, Using the Therascreen® KRAS RGQ PCR Kit, From Patients With Non-Small Cell Lung Cancer and Colorectal Cancer, Screened in Amgen's Clinical Trial (Protocol No. 20170543).
Brief Title: Clinical Performance Study Protocol for Therascreen® KRAS RGQ PCR Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QMAN-18-0181-1-001
Record Dates: First submitted 2022-04-01; First posted 2022-04-27 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Masking Description: Specimens from advanced NSCLC and CRC patient tumor samples, will be extracted and tested with the therascreen® KRAS RGQ PCR Kit. The sample KRAS G12C mutation status, if known by a previous testing method, will be blinded to device investigation site personnel at NeoGenomics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Performance Study Protocol for therascreen® KRAS RGQ PCR Kit (Other): The therascreen KRAS RGQ PCR Kit is a real-time qualitative PCR assay used on the Rotor-Gene Q MDx instrument for the detection of somatic G12C mutations in the human KRAS oncogene using DNA extracted from formalin fixed paraffin-embedded (FFPE) Colorectal Cancer (CRC) and Non-small Cell Lung Cancer (NSCLC) tissue. The therascreen KRAS RGQ PCR Kit is intended to aid in the identification of cancer patients who may be eligible for treatment with AMG 510.
  Interventions: Diagnostic Test: therascreen® KRAS RGQ PCR Kit

INTERVENTIONS:
Diagnostic Test: therascreen® KRAS RGQ PCR Kit — The primary objective is to utilize a clinical trial assay, the therascreen® KRAS RGQ PCR Kit, as a screening test in Phase 2 of Amgen clinical trial, in order to identify patients (with NSCLC and CRC) with KRAS G12C mutation positive tumors

SUMMARY:
An interventional, prospective clinical performance study protocol, for the testing of DNA extracted from tumor tissue biopsy samples, using the therascreen® KRAS RGQ PCR Kit, from patients with Non-Small Cell Lung Cancer and Colorectal Cancer, screened in Amgen's clinical trial (Protocol No. 20170543).

DETAILED DESCRIPTION:
This is an interventional, prospective clinical performance study protocol, for the testing of DNA extracted from tumor tissue biopsy samples (either core needle (NSCLC only) or excisional biopsies), obtained from patients with Non-Small Cell Lung Cancer (NSCLC) and Colorectal Cancer (CRC), using the therascreen® KRAS RGQ PCR Kit, (hereafter referred to as KRAS Kit).

Up to 280 patient tissue samples (from approximately 100 clinical study sites), obtained in the Amgen Clinical Protocol 20170543 study, will be tested using the KRAS Kit. The testing will be performed at the investigational device clinical testing site, NeoGenomics Laboratories, Inc., 7256 S. Sam Houston Pkwy W., Suite 300, Houston, Texas, 77085, USA.

The primary objective of the Amgen Clinical Study is to evaluate tumor objective response rate (ORR) assessed by MODIFIED RECIST 1.1 criteria of AMG 510 as a monotherapy in patients using the Clinical Trial Assay, therascreen® KRAS RGQ PCR Kit to assess whether to treat patients with KRAS G12C mutated advanced tumors (NSCLC and CRC).

The clinical data from the study will be used to determine the drug-device efficacy to support future regulatory submissions for the device-drug combination.

ELIGIBILITY:
Inclusion Criteria:

* All patients who provided consent (by signing and dating the Consent Form for Amgen Protocol No. 20170543), may be included in the device study.

Exclusion Criteria:

* Patients whose tumor tissue biopsy samples are not Clinical Trial Assay evaluable will be excluded from the study. Additionally, patients with samples identified for the study which have insufficient testing material will also be excluded, as will specimens which have undergone decalcification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
therascreen® KRAS RGQ PCR Kit | 5 business days
  therascreen® KRAS RGQ PCR Kit, as a screening test in Phase 2 of clinical trial (Protocol 20170543), in order to identify patients (with NSCLC and CRC) with KRAS G12C mutation positive tumors for inclusion in study (Protocol 20170543)

CONTACTS AND LOCATIONS:
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No